CLINICAL TRIAL: NCT05087862
Title: A Randomized Comparison Between Periarticular Infiltration of Local Anesthetics and Ultrasound-Guided Pericapsular Nerve Group Block for Total Hip Replacement
Brief Title: Periarticular Infiltration of Local Anesthetics Versus Pericapsular Nerve Group Block for Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, Assistant Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OAIC 1169/20
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain; Weakness, Muscle; Analgesia; Motor Activity
MeSH Terms: conditions — Pain, Postoperative; Muscle Weakness; Agnosia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective randomized comparison between two analgesic techniques
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular nerve group block (Active Comparator): Twenty milliliters of bupivacaine 0.5% (100 milligrams) with epinephrine 5 ug/mL will be deposited in the anterior aspect of the iliac bone between its periosteum and the tendon of the iliopsoas muscle. Additionally, ketorolac 30 mg will be administered intravenously.
  Interventions: Procedure: Ultrasound-guided pericapsular nerves group of the hip block
- Periarticular local anesthetic infiltration (Experimental): Sixty milliliters of 0.25% bupivacaine (150 milligrams), 5ug/mL epinephrine, and ketorolac 30 mg will be deposited at the periarticular level under direct vision during surgery. Fascia, subcutaneous tissues, and skin will also be infiltrated with part of the solution before wound closure.
  Interventions: Procedure: Pericapsular local anesthetic infiltration of the hip

INTERVENTIONS:
Procedure: Ultrasound-guided pericapsular nerves group of the hip block — After the ultrasound-guided insertion of a block needle at the level of the inguinal ligament, the needle will be advance into the plane between the iliac bone periosteum and the tendon of the iliopsoas muscle in order to inject 20 mL of adrenalized 0.5% bupivacaine.
  Arms: Pericapsular nerve group block
Procedure: Pericapsular local anesthetic infiltration of the hip — Intraoperatively, 60 mL of adrenalized 0.25% bupivacaine plus ketorolac 30 mg will be infiltrated by the surgeon.
  Arms: Periarticular local anesthetic infiltration

SUMMARY:
This randomized trial is set out to compare the postoperative strength preservation capacity of local infiltration anesthesia (LIA) and pericapsular nerve group (PENG) block after performing a primary total hip arthroplasty (THA).

The hypothesis is that LIA represents a superior alternative to PENG block in terms of strength preservation but providing effective analgesia during the first 24 postoperative hours after THA. Hence, the trial was designed as a superiority study hypothesizing a fivefold reduction in quadriceps paresis/paralysis at 3 hours.

DETAILED DESCRIPTION:
Patients who agree to participate in the protocol will be assigned to one group or another (LIA and PENG) through computationally generated block randomization. Outcome assessors blinded to randomization will perform all measurements.

All blocks, LIA or PENG, will be performed (or supervised) by one of the co-authors, an expert orthopedic surgeon or an expert anesthesiologist, respectively. Both blocks will be executed in the operating room, on the surgical table, under sedation, and with the barrier that separates the surgical field from the cranial area of the patient to keep the latter blind to the technique received.

All patients will undergo spinal anesthesia using 0.5% bupivacaine (10mg) plus 20 μg of fentanyl. Both groups will also receive tranexamic acid 1g intravenous (IV), ketoprofen 100mg IV, and acetaminophen 1gr IV. Propofol sedation guided with a targeted controlled infusion (TCI) model will be administered in order to obtain an adequate level of sedation.

All surgeries will be conducted by the same team of surgeons, performing a posterior approach technique in the lateral decubitus position.

In the recovery room, all patients will receive patient-controlled analgesia (morphine bolus = 1 mg; lockout interval = 8 minutes). On the surgical ward, all subjects will continue to receive acetaminophen (1 g per os every 6 hours), ketoprofen (100 mg per os every 8 hours) as well and patient-controlled analgesia (morphine bolus = 1 mg IV; lockout interval = 8 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 35 (kg/m2)

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 01.4 or prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* Allergy to local anesthetics (LAs) or morphine
* Pregnancy
* Prior surgery in the inguinal area of the corresponding surgical side
* Previous hip arthroplasty due to hip fracture
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Presence of quadriceps motor block (defined as paralysis or paresis) | 3 hours after post anesthesia care unit (PACU) arrival
  Quadriceps motor function will be tested with the patient lying on the bed and with the hip joint at 45º and the knee at 90º. The subject will be asked to extend the knee, first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).

SECONDARY OUTCOMES:
Presence of quadriceps motor block (defined as paralysis or paresis) | 6 hours after PACU arrival
  Quadriceps motor function will be tested with the patient lying on the bed and with the hip joint at 45º and the knee at 90º. The subject will be asked to extend the knee, first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).
Presence of quadriceps motor block (defined as paralysis or paresis) | 24 hours after PACU arrival
  Quadriceps motor function will be tested with the patient lying on the bed and with the hip joint at 45º and the knee at 90º. The subject will be asked to extend the knee, first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).
Hip adduction strength | 3 hours after PACU arrival
  Hip adduction will be evaluated by comparing it to baseline strength (i.e., prior to spinal anesthesia). A blood pressure cuff, inflated at 40 mmHg, will be inserted between the knees of the patient: the latter will then be instructed to squeeze the cuff as hard as possible and to sustain the effort. We will define hip adduction scores of 0, 1, and 2 points as decreases in strength of 0-20% (normal strength), 21-70% (paresis), and 71-90% (paralysis) compared to the baseline measurement, respectively.
Hip adduction strength | 6 hours after PACU arrival
  Hip adduction will be evaluated by comparing it to baseline strength (i.e., prior to spinal anesthesia). A blood pressure cuff, inflated at 40 mmHg, will be inserted between the knees of the patient: the latter will then be instructed to squeeze the cuff as hard as possible and to sustain the effort. We will define hip adduction scores of 0, 1, and 2 points as decreases in strength of 0-20% (normal strength), 21-70% (paresis), and 71-90% (paralysis) compared to the baseline measurement, respectively.
Hip adduction strength | 24 hours after PACU arrival
  Hip adduction will be evaluated by comparing it to baseline strength (i.e., prior to spinal anesthesia). A blood pressure cuff, inflated at 40 mmHg, will be inserted between the knees of the patient: the latter will then be instructed to squeeze the cuff as hard as possible and to sustain the effort. We will define hip adduction scores of 0, 1, and 2 points as decreases in strength of 0-20% (normal strength), 21-70% (paresis), and 71-90% (paralysis) compared to the baseline measurement, respectively.
Postoperative morphine consumption | 24 hours after PACU arrival
  Consumption of intravenous morphine (mg) registered by a patient-controlled analgesia device.
Postoperative morphine consumption | 48 hours after PACU arrival
  Consumption of intravenous morphine (mg) registered by a patient-controlled analgesia device.
Time until first morphine demand | 48 hours after PACU arrival
  Time (minutes) until first patient-controlled analgesia morphine demand.
Static and dynamic pain | 3 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 6 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 12 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 18 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 24 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Static and dynamic pain | 48 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Sensory block | 3 hours after PACU arrival
  Sensory block in the anterior, lateral and medial aspects of the mid-thigh. For each territory, blockade will be evaluated using a 3-point scale: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch)
Sensory block | 6 hours after PACU arrival
  Sensory block in the anterior, lateral and medial aspects of the mid-thigh. For each territory, blockade will be evaluated using a 3-point scale: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch)
Sensory block | 24 hours after PACU arrival
  Sensory block in the anterior, lateral and medial aspects of the mid-thigh. For each territory, blockade will be evaluated using a 3-point scale: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch)
Block/Infiltration-related complications | 1 hour after nerve block or local anesthetic infiltration
  Incidence of adverse events related to nerve block or local anesthetic infiltration (i.e. vascular puncture, local anesthetic systemic toxicity)
Postoperative opioid related side effects | 48 hours after PACU arrival
  Presence of postoperative nausea, vomiting, pruritus, urinary retention, respiratory depression.
Duration of surgery | 4 hours after skin incision
  Time between skin incision and closure (min)
Inability to perform physiotherapy due to motor block | 6 hours after PACU arrival
  Number of participants that cannot end the physiotherapy protocol programmed for the sixth hour after PACU arrival secondary to decreased strength in the operated limb.
Inability to perform physiotherapy due to motor block | Postoperative day 1
  Number of participants that cannot end the physiotherapy protocol programmed for the first postoperative day secondary to decreased strength in the operated limb.
Inability to perform physiotherapy due to motor block | Postoperative day 2
  Number of participants that cannot end the physiotherapy protocol programmed for the second postoperative day secondary to decreased strength in the operated limb.
Inability to perform physiotherapy due to pain | 6 hours after PACU arrival
  Number of participants that cannot end the physiotherapy protocol programmed for the sixth hour after PACU arrival secondary to pain in the operated limb.
Inability to perform physiotherapy due to pain | Postoperative day 1
  Number of participants that cannot end the physiotherapy protocol programmed for the first postoperative day secondary to pain in the operated limb.
Inability to perform physiotherapy due to pain | Postoperative day 2
  Number of participants that cannot end the physiotherapy protocol programmed for the second postoperative day secondary to pain in the operated limb.
Readiness to discharge | 4 days after surgery
  Days to be ready for discharge following physiotherapist criteria
Length of hospital stay | 7 days after surgery
  Length of hospital stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Julián Aliste, MD, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Wainwright TW, Gill M, McDonald DA, Middleton RG, Reed M, Sahota O, Yates P, Ljungqvist O. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Feb;91(1):3-19. doi: 10.1080/17453674.2019.1683790. Epub 2019 Oct 30. PMID 31663402
- [Background] Kuchalik J, Magnuson A, Lundin A, Gupta A. Local infiltration analgesia or femoral nerve block for postoperative pain management in patients undergoing total hip arthroplasty. A randomized, double-blind study. Scand J Pain. 2017 Jul;16:223-230. doi: 10.1016/j.sjpain.2017.05.002. Epub 2017 Jun 1. PMID 28850408
- [Background] Layera S, Saadawi M, Tran Q, Salinas FV. Motor-Sparing Peripheral Nerve Blocks for Shoulder, Knee, and Hip Surgery. Adv Anesth. 2020 Dec;38:189-207. doi: 10.1016/j.aan.2020.08.003. Epub 2020 Oct 1. No abstract available. PMID 34106834
- [Background] Husted C, Gromov K, Hansen HK, Troelsen A, Kristensen BB, Husted H. Outpatient total hip or knee arthroplasty in ambulatory surgery center versus arthroplasty ward: a randomized controlled trial. Acta Orthop. 2020 Feb;91(1):42-47. doi: 10.1080/17453674.2019.1686205. Epub 2019 Nov 4. PMID 31680610
- [Background] Bravo D, Layera S, Aliste J, Jara A, Fernandez D, Barrientos C, Wulf R, Munoz G, Finlayson RJ, Tran Q. Lumbar plexus block versus suprainguinal fascia iliaca block for total hip arthroplasty: A single-blinded, randomized trial. J Clin Anesth. 2020 Nov;66:109907. doi: 10.1016/j.jclinane.2020.109907. Epub 2020 Jun 2. PMID 32502775
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085
- [Background] Murphy TP, Byrne DP, Curtin P, Baker JF, Mulhall KJ. Can a periarticular levobupivacaine injection reduce postoperative opiate consumption during primary hip arthroplasty? Clin Orthop Relat Res. 2012 Apr;470(4):1151-7. doi: 10.1007/s11999-011-2108-3. Epub 2011 Sep 30. PMID 21960156
- [Derived] Bravo D, Aliste J, Layera S, Fernandez D, Erpel H, Aguilera G, Arancibia H, Barrientos C, Wulf R, Leon S, Branes J, Finlayson RJ, Tran Q. Randomized clinical trial comparing pericapsular nerve group (PENG) block and periarticular local anesthetic infiltration for total hip arthroplasty. Reg Anesth Pain Med. 2023 Oct;48(10):489-494. doi: 10.1136/rapm-2023-104332. Epub 2023 Feb 16. PMID 36797036